CLINICAL TRIAL: NCT03631810
Title: Contemporary Clinical Management Of Acute Pulmonary Embolism. The COPE Study
Brief Title: Contemporary Clinical Management Of Acute Pulmonary Embolism
Acronym: COPE
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Collaborators: University Of Perugia (Other)
Responsible Party: Sponsor
Other Study IDs: CRU_UniPg_2017
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2020-02

CONDITIONS: Acute Pulmonary Embolism
Keywords: Acute pulmonary embolism; International guidelines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute pulmonary embolism is a potentially life-threatening disease with short-term mortality ranges from less than 1% to more than 30% during the hospital stay. Recent guidelines recommend to tailor diagnosis hospitalization and acute treatment based on the estimated risk for short-term Death.

The assessment of the contemporary clinical management of patients with acute pulmonary embolism across different specialties would be of crucial value.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, multicenter study in patients with acute pulmonary embolism admitted to Cardiology, Emergency and Internal Medicine Departments in Italy.

The aim of the study is to assess contemporary management strategies in patients with acute pulmonary embolism in terms of diagnosis, risk stratification, hospitalization and treatment in Italy and assess

1. their association with in-hospital and 30-day mortality and
2. their adherence to current guidelines of the European Society of Cardiology (ESC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute, symptomatic acute pulmonary embolism
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

* refusal of informed consent
* participation in controlled trials on the management of patients with acute pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute symptomatic objectively diagnosed pulmonary embolism (first or recurrent).
Sampling Method: Non-Probability Sample
Enrollment: 5213 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
In-hospital death | 30 days
  In-hospital Death and Death at 30 days

SECONDARY OUTCOMES:
All cause Mortality and clinical worsening | 30 days
  Death or clinical deterioration at 30 days from the diagnosis of pulmonary embolism
Pulmonary embolism related mortality for and clinical worsening | 30 days
  Pulmonary embolism-related death or clinical deterioration at 30 days from the diagnosis of pulmonary embolismembolism
Adherence to guidelines | 30 days
  Adherence to current guidelines on the management of acute pulmonary embolism released by the ESC regarding diagnosis, risk stratification and treatment

CONTACTS AND LOCATIONS:
Locations (182):
- Italy (182):
  - Ospedale San Giovanni Di Dio - Uo Cardiologia E Utic, Agrigento, AG
  - Ospedali Riuniti - Sod Ps E Medicina D'Urgenza, Ancona, AN
  - Istituto Scientifico Inrca - Uo Cardiologia/Utic/Telecardiologia, Ancona, AN
  - Ospedale Madonna Del Soccorso - Medicina D'Urgenza, San Benedetto del Tronto, AP
  - Ospedale Civile Ss. Filippo E Nicola - Uosd Angiologia, Avezzano, AQ
  - Ospedale San Donato - Medicina Interna, Arezzo, AR
  - Ospedale Civile - Medicina Interna, Bibbiena, AR
  - Ospedale Valdichiana Santa Margherita - Uos Cardiologia E Hdu, Cortona, AR
  - Osp. Valdarno 'S. Maria Della Gruccia' - Medicina Interna, Montevarchi, AR
  - Ospedale Cardinal Massaia - Medicina A, Asti, AT
  - Po Sant'Ottone Frangipane - Medicina Generale, Ariano Irpino, AV
  - Aorn San Giuseppe Moscati - Medicina Interna, Avellino, AV
  - Ospedale Di Venere - U.O.C. Di Cardiologia, Bari, BA
  - Ospedale San Paolo - Cardiologia-Utic, Bari, BA
  - Ospedale Policlinico - U.O. Cardiologia Universitaria, Bari, BA
  - Ospedale Policlinico - U.O. Di Cardiologia Ospedaliera, Bari, BA
  - Asst Papa Giovanni Xxiii - Centro Eas, Bergamo, BG
  - Asst Papa Giovanni Xxiii - Divisione Di Medicina Interna, Bergamo, BG
  - Iob - Policlinico San Marco - U.O. Cardiologia, Osio Sotto, BG
  - Ospedali Treviglio-Caravaggio - Cardiologia, Treviglio, BG
  - Ospedale Policlinico S. Orsola-Malpighi - Uoc Medicina D'Urgenza E Pronto Soccorso, Bologna, BO
  - Ospedale Maggiore - Medicina Interna A, Bologna, BO
  - Ospedale Nuovo S. Maria Della Scaletta - Medicina D'Urgenza E Pronto Soccorso, Imola, BO
  - Ospedale Perrino - U.O.C. Di Cardiologia, Brindisi, BR
  - Istituto Osped. Fondazione Poliambulanza - Unita' Operativa Di Cardiologia, Brescia, BS
  - Ospedale Civile 'La Memoria' - U.O. Di Cardiologia, Gavardo, BS
  - Osp. Andria Canosa - Po Andria - Cardiologia - Utic, Andria, BT
  - Az. Ospedaliera S. Anna E S. Sebastiano - Medicina D'Urgenza, Caserta, CE
  - Pineta Grande Hospital - Medicina D'Urgenza, Castel Volturno, CE
  - Ospedale 'Renzetti' - Medicina Interna, Lanciano, CH
  - Azienda Ospedaliera Santa Croce E Carle - Divisione Di Medicina Interna, Cuneo, CN
  - Ospedale Maggiore Ss. Annunziata - Medicina E Chirurgia D'Urgenza, Savigliano, CN
  - Ospedale S. Anna - U.O.C. Di Cardiologia, San Fermo della Battaglia, CO
  - Ospedale Civile Oglio Po - Medicina Generale, Casalmaggiore, CR
  - Ospedale Di Cremona - Medicina Interna, Cremona, CR
  - Ospedale Annunziata - Uoc Cardiologia, Cosenza, CS
  - P.O. Garibaldi-Nesima - U.O.C. Di Cardiologia, Catania, CT
  - P.O. Garibaldi Centro - U.O.C. Cardiologia, Catania, CT
  - Policlinico Catania Po G. Rodolico - Cardiologia Utic, Catania, CT
  - Azienda Ospedaliera Cannizzaro - Medicina Interna, Catania, CT
  - Azienda Ospedaliera Cannizzaro - Uoc Cardiologia Con Utic Ed Emodinamica, Catania, CT
  - P.O. Garibaldi Centro - Medicina Interna Area Critica, Catania, CT
  - Ospedale Civile Pugliese - Utic-Emodinamica E Card. Interventistica, Catanzaro, CZ
  - Ospedale Giovanni Paolo Ii - U.O. Cardiologia E Utic, Lamezia Terme, CZ
  - Ospedale G.B. Morgagni - L. Pierantoni - U.O. Cardiologia, Forlì, FC
  - Ospedale G.B. Morgagni - L. Pierantoni - U.O. Medicina D'Urgenza-Pronto Soccorso, Forlì, FC
  - Ospedali Riuniti - S.C. Di Cardiologia Univ.-Utic, Foggia, FG
  - Presidio Ospedaliero T. Masselli Mascia - S.C. Cardiologia - Utic - Riabil. Card., San Severo, FG
  - Ospedale Santa Maria Annunziata - Dea, Bagno a Ripoli, FI
  - Ospedale Civile San Giuseppe - Medicina D'Urgenza, Empoli, FI
  - Ospedale Civile San Giuseppe - Medicina Interna Ii, Empoli, FI
  - Presidio Ospedaliero Serristori - Medicina Interna E D'Urgenza, Figline Valdarno, FI
  - Ospedale Santa Maria Nuova - Medicina A2, Florence, FI
  - Ospedale San Giovanni Di Dio - Medicina Interna, Florence, FI
  - Ospedale Civile Augusto Murri - Medicina Interna, Fermo, FM
  - Ospedale Civile Augusto Murri - U.O. Cardiologia, Fermo, FM
  - Ospedale Fabrizio Spaziani - Cardiologia-Utic, Frosinone, FR
  - E.O. Ospedali Galliera - Medicina Interna, Genova, GE
  - E.O. Ospedali Galliera - S. C. Cardiologia, Genova, GE
  - Ospedale Policlinico San Martino - Medicina D'Urgenza 1, Genova, GE
  - Ospedale Policlinico San Martino - Unita' Operativa Cardiologia, Genova, GE
  - Ospedale Padre Antero Micone - Sc Cardiologia - Utic, Genova, GE
  - Ospedale Della Misericordia - Pronto Soccorso, Grosseto, GR
  - Ospedale S. Andrea - Alta Maremma - Divisione Di Medicina, Massa Marittima, GR
  - Presidio Ospedaliero - U.O. Cardiologia, Sanremo, IM
  - Ospedale Alessandro Manzoni - S.C. Di Cardiologia, Lecco, LC
  - Presidio Ospedaliero F. Ferrari - Cardiologia - Utic, Casarano, LE
  - Ospedale Civile Sacro Cuore Di Gesu' - Uo Cardiologia Utic, Gallipoli, LE
  - Ospedale Civile Bassa Val Di Cecina - Medicina Generale, Cecina, LI
  - Ospedali Riuniti - Medicina Generale, Livorno, LI
  - Ospedali Riuniti - Pronto Soccorso E Medicina D'Urgenza, Livorno, LI
  - Ospedale Villamarina - Medicina Generale, Piombino, LI
  - Presidio Ospedaliero Di Lodi - Medicina Generale, Lodi, LO
  - Nuovo Ospedale Versilia - Medicina Generale, Lido di Camaiore, LU
  - Nuovo Ospedale Versilia - Pronto Soccorso, Lido di Camaiore, LU
  - Ospedale San Gerardo - U.O. Cardiologia-Utic, Monza, MB
  - Policlinico Di Monza - Uo Cardiol. Clinica E Scompenso Cardiaco, Monza, MB
  - Ospedale Civile - Medicina Generale, Legnano, MI
  - Ospedale Civile Fornaroli - Medicina Interna, Magenta, MI
  - Ospedale Maggiore Policlinico - Pronto Soccorso E Medicina D'Urgenza, Milan, MI
  - Multimedica Ospedale San Giuseppe - Pneumologia, Milan, MI
  - Centro Cardiologico Monzino - Terapia Intensiva Cardiologica (Utic), Milan, MI
  - Ospedale San Luca - Istituto Auxologico - U.O. Cardiologia, Milan, MI
  - Ospedale San Carlo Borromeo - Cardiologia-Ucc, Milan, MI
  - Ospedale San Carlo Borromeo - Pronto Soccorso E Medicina D'Urgenza, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Cardiologia 1 - Emodinamica, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Medicina D'Urgenza E Pronto Soccorso, Milan, MI
  - Asst Ospedale Metropolitano Niguarda - Medicina Interna 1, Milan, MI
  - Irccs Policlinico Multimedica - Uo Di Cardiologia, Sesto San Giovanni, MI
  - Ospedale Madonna Delle Grazie - Pronto Soccorso Tsi, Matera, Mount
  - Ospedale Madonna Delle Grazie - U.O. Cardiologia Utic, Matera, Mount
  - Ospedale Policlinico - Pronto Soccorso, Modena, MO
  - Ospedale Policlinico - Uo Cardiologia, Modena, MO
  - Ospedale Civile Di Baggiovara - Medicina D'Urgenza E Pronto Soccorso, Modena, MO
  - Presidio Ospedaliero - Divisione Di Medicina Generale, Pavullo nel Frignano, MO
  - Ospedale Di Sassuolo - Medicina D'Urgenza, Sassuolo, MO
  - Ospedale Di Sassuolo - Medicina Interna, Sassuolo, MO
  - Ospedale Civile - Uo Pronto Soccorso, Vignola, MO
  - Ospedale San Francesco - Cardiologia - Utic, Nuoro, NU
  - Osp. Buccheri La Ferla Fatebenefratelli - Dip. Emergenza, Accettaz. E Dei Servizi, Palermo, PA
  - Aor Villa Sofia-Cervello Po Villa Sofia - U.O.C. Cardiologia E Utic - Villa Sofia, Palermo, PA
  - Ospedale Di Cittadella - U.O. Cardiologia, Cittadella, PD
  - Ospedale Civile Dello Spirito Santo - Uo Geriatria, Pescara, PE
  - Presidio Ospedaliero Citta' Di Castello - Medicina Interna, Città di Castello, PG
  - Presidio Ospedaliero Citta' Di Castello - U.O. Di Cardiologia, Città di Castello, PG
  - Azienda Ospedaliera Di Perugia - Medicina Interna Vascolare E D'Urgenza, Perugia, PG
  - Nuovo Ospedale Media Valle Del Tevere - Divisione Di Medicina Interna, Todi, PG
  - Ospedale Generale Provinciale Lotti - U.O. Malattie Cardiovascolari, Pontedera, PI
  - Ospedale Di Pordenone - Ps E Medicina D'Urgenza, Pordenone, PN
  - Ospedale Di Pordenone - S.O.C. Cardiologia, Pordenone, PN
  - Ospedale Della Val Di Nievole - U. O. Cardiologia - Utic, Pescia, Point
  - Ospedale Santo Stefano - Pronto Soccorso E Medicina D'Urgenza, Prato, PO
  - Ospedale Civile - Ps E Medicina D'Urgenza, Fidenza, PR
  - Presidio Ospedaliero San Salvatore - Cardiologia E Utic, Pesaro, PU
  - Fondazione Irccs Policlinico San Matteo - Pronto Soccorso, Pavia, PV
  - Ospedale S. Giovanni Di Dio - U.O. Cardiologia E Utic, Melfi, PZ
  - Azienda Ospedaliera San Carlo - Ssd Utic, Potenza, PZ
  - Azienda Ospedaliera San Carlo - Uoc Ps Accettazione Medicina D'Urgenza, Potenza, PZ
  - Ospedale Per Gli Infermi - Pronto Soccorso, Faenza, RA
  - Ospedale Civile Santa Maria Delle Croci - Pronto Soccorso E Medicina D'Urgenza, Ravenna, RA
  - Ao Bianchi Melacrino Morelli- Po Riuniti - Divisione Di Cardiologia, Reggio Calabria, RC
  - Arcispedale Santa Maria Nuova - Medicina Cardiovascolare, Reggio Emilia, RE
  - Arcispedale Santa Maria Nuova - Medicina D'Urgenza E Pronto Soccorso, Reggio Emilia, RE
  - Ospedale Magati - Divisione Di Medicina-Area Internistica, Scandiano, RE
  - Ospedale Riccardo Guzzardi - U.O.C. Di Cardiologia-Utic, Vittoria, RG
  - P.O. San Filippo Neri - Asl Roma 1 - Uoc Cardiologia E Utic, Roma, RM
  - Ospedale San Camillo - Cardiologia 2 (Ex Cardio 3), Roma, RM
  - Ospedale San Camillo - Medicina D'Urgenza E Cure Differenziate, Roma, RM
  - Ospedale Sandro Pertini - Medicina D'Urgenza, Roma, RM
  - Policlinico Umberto Primo - Cardiologia B - Cardiologia E Angiologia, Roma, RM
  - Policlinico Casilino - U.O. Cardiologia, Roma, RM
  - Ao San Giovanni Addolorata - Uoc Ps-Breve Osservazione, Roma, RM
  - Ospedale Fatebenefratelli - Medicina Interna, Roma, RM
  - Ospedale Sant'Andrea Di Roma - U.O.C. Cardiologia, Roma, RM
  - Ospedale Santo Spirito - U.O.C. Di Cardiologia, Roma, RM
  - Ospedale Infermi - U.O. Cardiologia, Rimini, RN
  - Ospedale Santa Maria Della Misericordia - U.O.C. Cardiologia, Rovigo, RO
  - Ospedale Santa Maria Della Misericordia - Uoc Medicina Interna - Angiologia, Rovigo, RO
  - Ospedale Dell'Alta Val D'Elsa - Uosd Cardiologia-Utic, Poggibonsi, SI
  - Aou Senese Ospedale S. Maria Alle Scotte - Uoc Medicina Interna 2, Siena, SI
  - Ospedale S. Andrea - Medicina Interna, La Spezia, SP
  - Ospedale E. Muscatello - U.O. Di Cardiologia - Utic, Augusta, SR
  - Ospedale Umberto I - Div. Di Medicina - Centro Ipertensione, Syracuse, SR
  - Ospedale Ss. Annunziata - Pronto Soccorso E Medicina D'Urgenza, Sassari, SS
  - Ospedale San Paolo - Medicina Interna E Cure Intermedie, Savona, SV
  - Ospedale Civile M. Giannuzzi - Cardiologia E Utic, Manduria, TA
  - Ospedale Civile G. Mazzini - Uoc Pronto Soccorso, Teramo, TE
  - Ospedale Santa Maria Del Carmine - Medicina Interna, Rovereto, TN
  - Ospedale Santa Chiara - Medicina Interna I, Trento, TN
  - Ospedale Civile San Lazzaro - Medicina Generale, Alba, TO
  - Ospedale Maggiore - Sc Medicina Interna, Chieri, TO
  - Ospedale Civile E. Agnelli - Medicina-Chirurgia Accettazione-Urgenza, Pinerolo, TO
  - Ospedale Degli Infermi - Medicina Generale, Rivoli, TO
  - Ospedale Maria Vittoria - U.O. Cardiologia, Torino, TO
  - Ospedale Humanitas Gradenigo - Medicina E Chirurgia D'Urgenza, Torino, TO
  - Ospedale Civile Sant'Antonio Abate - U.O.C. Di Cardiologia E Utic, Erice, TP
  - Ospedali Riuniti - Osp. Cattinara - Medicina D'Urgenza E Ps, Trieste, TS
  - Ospedali Riuniti - Osp. Cattinara - S.O.C. Cardiologia, Trieste, TS
  - Stabilimento Ospedaliero Di Castelfranco - Uoc Angiologia, Castelfranco Veneto, TV
  - Ospedale San Valentino - Divisione Di Medicina Interna, Montebelluna, TV
  - Ospedale Ca' Foncello - Pronto Soccorso Medicina D'Urgenza, Treviso, TV
  - Pou Santa Maria Della Misericordia - Pronto Soccorso Medicina D'Urgenza, Udine, UD
  - Ospedale Di Luino - Medicina Generale, Luino, VA
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno, VA
  - Ospedale Di Circolo E Fondazione Macchi - Geriatria, Varese, VA
  - Ospedale Di Circolo E Fondazione Macchi - Medicina Generale I, Varese, VA
  - Ospedale Sant'Andrea - Medicina Interna, Vercelli, VC
  - Ospedale Civile - Medicina Interna, Arzignano, VI
  - Ospedale Civile - U.O.C. Cardiologia, Arzignano, VI
  - Ospedale San Bassiano - Sc Di Medicina Interna, Bassano del Grappa, VI
  - Ospedale Civile - Medicina Generale 2, Noventa Vicentina, VI
  - Ospedale Civile San Bortolo - U.O.C. Cardiologia, Vicenza, VI
  - Ospedale G. Fracastoro - U.O.C. Di Cardiologia, San Bonifacio, VR
  - Aoui Di Verona - Medicina Gen. Malattie Aterotrombotiche, Verona, VR
  - Ospedale Belcolle - Medicina Generale, Viterbo, VT
  - Ospedale Civile G. Jazzolino - Medicina D'Urgenza, Vibo Valentia, VV
  - Ospedale Buon Consiglio Fatebenefratelli - Struttura Complessa Di Medicina, Napoli
  - Aorn Cardarelli - Medicina D'Urgenza, Napoli
  - Aou Federico Ii - Uoc Cardiologia E Utic, Napoli
  - Aou Maggiore Della Carita' - Cardiologia Ii, Novara
  - Ospedale Della Val Di Nievole - Medicina Generale, Pescia
  - Ospedale Santa Maria Delle Grazie - U.O. Cardiologia - Utic, Pozzuoli

REFERENCES:
- [Derived] Becattini C, Agnelli G, Diamanti M, Maggioni AP, Vanni S, Dentali F, Enea I, Bortolotti P, De Vecchi M, Artusi N, Picariello C, Nitti C, Lucci D, Gulizia MM; COPE Investigators. Contemporary anticoagulant treatment strategies in patients with acute pulmonary embolism at different risk for death. Vascul Pharmacol. 2023 Dec;153:107245. doi: 10.1016/j.vph.2023.107245. Epub 2023 Nov 25. PMID 38013135
- [Derived] Becattini C, Cimini LA, Bassanelli G, Maggioni AP, Pomero F, Lobascio I, Enea I, Pomata DP, Ruggieri MP, Zalunardo B, Novelli A, Di Fusco SA, Triggiani M, Marzolo M, Fioravanti C, Agnelli G, Gonzini L, Gulizia MM; COPE Investigators. Acute pulmonary embolism and cancer: findings from the COPE study. Clin Res Cardiol. 2024 Feb;113(2):288-300. doi: 10.1007/s00392-023-02323-z. Epub 2023 Nov 15. PMID 37966670
- [Derived] Becattini C, Agnelli G, Maggioni AP, Dentali F, Fabbri A, Enea I, Pomero F, Ruggieri MP, di Lenarda A, Cimini LA, Pepe G, Cozzio S, Lucci D, Gulizia MM; COPE Investigators. Contemporary Management and Clinical Course of Acute Pulmonary Embolism: The COPE Study. Thromb Haemost. 2023 Jun;123(6):613-626. doi: 10.1055/a-2031-3859. Epub 2023 Feb 9. PMID 36758612
- [Derived] Becattini C, Agnelli G, Maggioni AP, Dentali F, Fabbri A, Enea I, Pomero F, Ruggieri MP, Di Lenarda A, Gulizia M. Contemporary clinical management of acute pulmonary embolism: the COPE study. Intern Emerg Med. 2022 Apr;17(3):715-723. doi: 10.1007/s11739-021-02855-0. Epub 2022 Jan 4. PMID 34982399